CLINICAL TRIAL: NCT03212469
Title: A Phase I/II Study Evaluating the Safety and Clinical Activity of Anti-PDL1 (Durvalumab [MEDI4736]) + Anti CTLA-4 (Tremelimumab) Antibodies Administrated in Combination With Stereotactic Body Radiotherapy (SBRT) in Patients With Metastatic Squamous Cell Carcinoma of Head and Neck, Lung, Oesophageus, Cervix, Vagina,Vulva or Anus
Brief Title: A Trial of Durvalumab and Tremelimumab in Combination With SBRT in Patients With Metastatic Cancer
Acronym: ABIMMUNE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-514920-18-00; 2016/2454 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2017-01-31; First posted 2017-07-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Lung Cancer; Oesophageal Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lung Neoplasms; Esophageal Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: The study is an open label, multicentric, Phase I/II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with head and neck squamous cell carcinoma (Experimental)
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: SBRT
- Patients lung cancer (Experimental)
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: SBRT
- Patients with oesophagus cancer (Experimental)
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: SBRT

INTERVENTIONS:
Drug: Durvalumab — Preliminary steps : Safety Runs Safety run of the dual combination Durvalumab as single agent at the selected dose of 1500mg, every 4 weeks (Q4W) from C1D1 up to 13 doses
  Safety run of the triple combination:
  Durvalumab at 1500mg every 4 weeks (Q4W) from C1D1 up to 13 doses,
  Efficacy step
  * Durvalumab Q4W + Tremelimumab Q4W for up to 4 doses at the DL defined in safety runs, in conjunction with
  * SBRT at C1D15, then
  * Durvalumab Q4W alone for up to 9 additional doses
Drug: Tremelimumab — Preliminary steps : Safety Runs
  Safety run of the triple combination:
  Tremelimumab at 75mg/Q4W for up to 4 doses
  Efficacy step
  * Durvalumab Q4W + Tremelimumab Q4W for up to 4 doses at the DL defined in safety runs, in conjunction with
  * SBRT at C1D15, then
  * Durvalumab Q4W alone for up to 9 additional doses
Radiation: SBRT — Preliminary steps : Safety Runs
  Safety run of the dual combination:
  SBRT at C1D15.
  Safety run of the triple combination:
  SBRT at C1D15.
  Efficacy step
  * Durvalumab Q4W + Tremelimumab Q4W for up to 4 doses at the DL defined in safety runs, in conjunction with
  * SBRT at C1D15, then
  * Durvalumab Q4W alone for up to 9 additional doses

SUMMARY:
The study is an open label, multicentric, Phase I/II trial aiming to evaluate the safety, the clinical activity and abscopal anti-tumor effects of a therapeutic strategy associating Durvalumab in conjunction with SBRT or Durvalumab + Tremelimumab in conjunction with SBRT in patients with metastatic squamous cell carcinoma of head and neck, lung, or esophagus.

ELIGIBILITY:
Inclusion Criteria:

I1. Male or Female patients ≥18 years of age or older.

I2. Histologically or cytologically proven metastatic squamous cell carcinoma (from head and neck, oesophagus, lung, cervix, vagina, vulva or anus) with the following features:

* Previously treated with at least one prior regimen (chemotherapy, signal transduction inhibitors or radiotherapy)
* To be treated with radiotherapy at primary tumor site or metastatic site or menacing metastatic site.
* The sites of metastases allowed are: soft tissue, peripheral lung, and liver.
* Patients with brain and bone metastasis to be treated with radiotherapy are not allowed. Patients with asymptomatic brain metastasis can be included.
* The total tumor volume to be irradiated must not exceed 400 cc.

I3. At least one tumor lesion must be accessible to radiation therapy and at least another tumor site can be spared from radiation therapy (unirradiated site).

I4. At least one unirradiated and one irradiated tumor site must be accessible to tumor biopsy.

I5. Known availability of an archived block

I6. The irradiated and unirradiated tumor sites must be measurable as per RECIST 1.1

I7. Patients must have no history of previous radiation therapy within the body area to be irradiated.

I8. Minimal wash-out periods from previous treatments to C1D1 must be

* Any investigational agent > 4 weeks
* Bevacizumab > 6 weeks
* Chemotherapy > 4 weeks
* TKI > 4 weeks
* RANK ligand agonists > 6 weeks
* Immunosuppressive medication > 28 days, with the exceptions of intranasal, topical, and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceeding 10 mg/day of prednisone, or an equivalent corticosteroid
* Live attenuated vaccination > 30 days

I9. WHO 0-1, Performance Status ECOG of 0-1

I10. Patients must have adequate organ function defined as follows:

* Absolute neutrophil count of ≥ 1500/mm3,
* Platelet count≥ 100,000/mm3,
* Hemoglobin > 9 g/dL,
* Bilirubin ≤ 1.5 times the institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* Serum ALT and AST ≤2.5 ULN (or if liver metastases are present must be ≤ 5x ULN)
* Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (see formula in section 4.1).

I11. Patients must be free of significant comorbid conditions that would preclude safe administration or completion of protocol therapy.

I12. Female patients must either be of non-reproductive potential (ie, postmenopausal ≥ 12 months with no menses without an alternative medical cause OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry (within 72 hours before study drug start).

I13. Fertile men with a female partner of childbearing potential must agree to use male condom plus spermicide and childbearing potential women must have agreed to use at least one highly effective contraceptive method during treatment on this trial and for up to 180 days after the last of dose of Durvalumab + Tremelimumab or 90 days after the last dose of Durvalumab monotherapy, whichever is the longer period.

I14. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.

I15. Patients must be affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

E1. Any situation where the irradiation of the target site would imply reirradiation of a formerly irradiated tumor site.

E2. Patients with any concurrent severe and/or uncontrolled disease which could compromise participation in the study including:

* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Active or prior documented autoimmune disease within the past 2 years. Of note, patient with vitiligo, Grave's disease or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Patients with type 1 diabetes or hypothyroidism stable under treatment or not requiring systemic treatment are eligible.
* Active or prior documented inflammatory bowel disease (eg Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* Severe chronic or acute infection such as chronic HBV, HCV and HIV1, 2 infection, active tuberculosis infection
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity or active non-infectious pneumonitis
* History of allogenic organ transplant
* Uncontrolled diabetes,
* Prior history of active bleeding diathesis or patients taking an oral vitamin K antagonist (except low-dose Coumadin (warfarin sodium))
* Symptomatic congestive heart failure,
* Uncontrolled hypertension,
* Unstable angina pectoris
* Cardiac arrhythmia
* Active peptic ulcer disease or gastritis,
* Any psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the sponsor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Patients with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Chronic treatment with corticosteroids or another immunosuppressant

E3. Patients with tumors that invade major vessels, as shown unequivocally by imaging studies

E4. Patients with central lung metastasis (i.e within 2 cm from hilum) that are cavitary as shown unequivocally by imaging studies

E5. Patients with a history of gross hemoptysis (bright red blood of 1/2 teaspoon or more per episode of coughing) ≤ 3 months prior enrolment

E6. Major surgery within the last 4 weeks prior to entering the study

E7. Persisting significant toxicities related to prior treatments i.e. ≥ Grade 2 AE according to CTCAE V4.03 except alopecia and biological values defined in inclusion criteria I10.

E8. Current or planned use of forbidden concomitant medications :

* Any investigational anticancer therapy not specified in this protocol
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for noncancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
* Immunosuppressive medications including, but not limited to systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent, methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications for the management of investigational product-related AEs or in subjects with contrast allergies is acceptable. In addition, use of topical, inhaled and intranasal corticosteroids is permitted.
* Live attenuated vaccines within 90 days of Durvalumab dosing or within 180 days of Durvalumab and Tremelimumab dosing. Inactivated vaccines, such as the injectable influenza vaccine, are authorized.

E9. Any prior Grade ≥ 3 irAE while receiving previous immunotherapy agent or any unresolved irAE > Grade 1.

E10. Prior exposure to any anti-PD-1 or anti-PD-L1 or anti-CTLA4 antibody.

E11. Known allergy or hypersensitivity to humanized antibodies.

E12. Pregnant or breastfeeding women.

E13. Persons deprived of their freedom or under guardianship, or for whom it would be impossible to undergo the medical follow-up required by the trial, for geographic, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Approximately 8 weeks
  Event possibly related to study drugs and fulfills any one of the following criteria using CTCAE Version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEUTSCH, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided